CLINICAL TRIAL: NCT04912375
Title: Executive Function, Reactivity to Cues of Food Consumption: a Cohort Study in Young Adults
Brief Title: Decision-making for Food Consumption in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021effood
Record Dates: First submitted 2021-05-27; First posted 2021-06-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low EF with priming (Experimental): Participants will be first stratified by their Executive function (EF). In this arm, participants have low EF. They will play a puzzle task that will ask participants to take 5 min to search Chinese words for meaningful statements. Each statement represents an implicit goal of healthy eating.
  Interventions: Behavioral: Priming intervention
- Low EF without priming (No Intervention): Participants will be first stratified by their Executive function (EF). In this arm, participants have low EF. They will play a similar puzzle task but the statements they searched are neutral.
- High EF with priming (Experimental): Participants will be first stratified by their Executive function (EF). In this arm, participants have high EF. They will play a puzzle task that will ask participants to take 5 min to search Chinese words for meaningful statements. Each statement represents an implicit goal of healthy eating.
  Interventions: Behavioral: Priming intervention
- High EF without priming (No Intervention): Participants will be first stratified by their Executive function (EF). In this arm, participants have high EF. They will play a similar puzzle task but the statements they searched are neutral.

INTERVENTIONS:
Behavioral: Priming intervention — The pilot RCT will ask participants to complete a simple word-searching exercise as a goal-priming of healthy eating and can be completed in 5 min.
  Arms: High EF with priming; Low EF with priming

SUMMARY:
Background: Experimental and cross-sectional evidence suggests that poor executive function can lead to heightened reactivity to food cues and perceived greater reward of unhealthy but palatable foods and subsequently lead to overeating or clinical eating disorders. This may be an important reason for the increasing trend of obesity in our society.

Aims: This study will investigate the interrelationships among executive function, reactivity to food-related cues and eating style in young adults. In addition, this study will examine the influence of food environment and stress on reactivity to food-related cues and executive function and how executive function and reactivity to food-related cues would influence health risky behaviours in young adults. We will also conduct a pilot randomized control trial (RCT) to develop the culturally specific goal priming intervention for the Chinese adults and test its effect on decision-making for food choice among adults with low executive function.

Design and subjects: This will be a three-wave cohort study in young adults who are recruited in their final-year of first post-secondary education and follow-up at six months and 12 months after their graduation. For the pilot RCT, a 2 (low vs. high executive function) x 2 (with vs. without goal priming intervention) will be used to test the effect of goal priming intervention on food choice. The goal priming intervention will be 5-min word-searching task to prime goals of healthy eating.

Main outcome measures: Participants will be invited to complete a series on computerized tasks and other assessments online in each wave to assess their executive function, risk taking propensity, reactivity to food-related cues, perceived stress, exposure to food-related cues, eating style and other health-related behaviours. Structural equation modelling will be used to test the interrelationships among executive function, reactivity to food-related cues and eating style, among exposure to food-related cues, perceived stress and reactivity to food-related cues, and among executive function, reactivity to food-related cues, risk taking and adoption of health-related behaviours. For the pilot RCT, the effect of intervention on tendency of choosing healthy and low-calorie foods will be evaluated using logistic regression model with level of executive function and goal-priming intervention as the main between-group factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who can speak Chinese or Mandarin
* Aged between 18 and 30 years

Exclusion Criteria:

* Having cognitive difficulties to understand the study instruments
* Having a physical or medical condition that requires certain food or dietary restrictions
* Having been diagnosed with any pathogenic eating disorders
* Participants whose subject is related to psychology

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
The effect of goal priming intervention on food choice | Immediately after participants completing the tasks
  The name of measure: participants' tendency to choose different categories of foods
  Measurement tool: the force food choice task
  * The force food choice task evaluates participants' 'wanting' of foods with tempting cues. ("if you had to make a choice, which food would you most want to eat now?")
  * Software: Survey responses and test data were recorded in Inquisit via the web or lab-based service.
  Unit of measure: the frequency of food selections

CONTACTS AND LOCATIONS:
Overall Officials: Qiuyan Liao, PhD, Principal Investigator — School of Public Health, University of Hong Kong
Locations (1):
- University of Hong Kong School of Public Health, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author upon reasonable request.